CLINICAL TRIAL: NCT00546052
Title: 52 Week Study to Evaluate the Effects of LOSARTAN 50 mg, 100 mg, 100/12.5 mg HCTZ, 100/25 mg HCTZ on Metabolic Parameters, Blood Pressure and Safety in Hypertensive Patients With Metabolic Syndrome
Brief Title: A 52 Week Study to Evaluate the Effects of Losartan With or Without HCTZ on Plasma Glucose, Metabolic Parameters, Blood Pressure in Hypertensive Patients With Metabolic Syndrome (0954A-331)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0954A-331; MK0954A-331; 2007_030
Record Dates: First submitted 2007-10-17; First posted 2007-10-18 (Estimated); Results first posted 2009-06-23 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2022-02

CONDITIONS: Hypertension; Metabolic Disorder
MeSH Terms: conditions — Hypertension; Metabolic Diseases | interventions — hydrochlorothiazide, losartan drug combination; Losartan

ARMS (1):
- 1 (Experimental): Losartan (MK0954) / Losartan + HCTZ (MK0954A)
  Interventions: Drug: losartan potassium (+) hydrochlorothiazide

INTERVENTIONS:
Drug: losartan potassium (+) hydrochlorothiazide — All patients received Losartan 50mg at Visit 2 titrated to Losartan 100mg (if target BP not achieved) titrated to Losartan 100mg + HCTZ 12.5mg (if necessary) up to Losartan 100mg + HCTZ 25mg. Duration of treatment was one year.
  Other Names: Cozaar/Hyzaar

SUMMARY:
To determine if a one year treatment Losartan with or without HCTZ at different dosages have an effect on metabolic parameters in patients with hypertension and the metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* An Adult Patient (At Least 18 Years Of Age) With A Clinical Identification Of The Metabolic Syndrome Using The IDF Definition:

  * abdominal (central) obesity as defined by the waist circumference in men of > 102 cm and women of > 88 cm or a BMI equal or greater than 30 kg/m2

and untreated hypertension with bp equal or greater than 140/90 mm Hg but bp < 180/110 mm Hg

or a patient receiving one or two antihypertensive agent(s) (diuretics, ace inhibitors, angiotensin ii receptor blockers, calcium channel blockers and beta-blockers will need to be discontinued) and whose blood pressure is not controlled:

* bp equal or greater than 140/90 mm Hg but equal or less than 160/100 mm Hg

or a patient whose hypertension is controlled (< 140/90 mm hg) with a single anti-hypertensive agent (diuretics, ace inhibitors, and angiotensin II receptor blockers, calcium channel blockers and beta-blockers will need to be discontinued) but who is unsatisfied or experiencing side effects warranting a discontinuation of the previous treatment and at one of the following:

* Fasting plasma glucose equal or greater than 5.6 mmol/L and < 7.0 mmol/L
* Triglycerides > 1.7 mmol/L or specific treatment for this lipid abnormality
* HDL-c in men < 0.9 mmol/L and in women < 1.1 mmol/L or specific treatment for this lipid abnormality

Exclusion Criteria:

* A Patient With A Diagnosis Of Type II Diabetes Defined As Fasting Blood Glucose Level Equal Or Greater Than 7.0 Mmol/L Or A 2hpg In A 75-G OGTT Equal Or Greater Than 11.1 Mol/L Or Using Any Anti-Hyperglycemic Agents
* Known Secondary Hypertension Of Any Aetiology (E.G., Uncorrected Renal Artery Stenosis, Malignant Hypertension, Or Hypertensive Encephalopathy)
* Patient Intolerant To Any Component Of Losartan 50 Mg / Losartan 100 Mg / Losartan 100 Mg + Hctz 12.5 Mg / Losartan 100 Mg + Hctz 25 Mg Or With A Documented History Of Angioedema
* Patient With Confirmed Clinically Significant Renal Or Hepatic Dysfunction And/Or Electrolyte Imbalance On The Basis Of The Case History Or A Recent Laboratory Test (Serum Creatinine > 130 Mmol/L Or Creatinine Clearance < 45 Ml/Min, Ast > 2 Times Above The Normal Range, Alt > 2 Times Above The Normal Range, Serum Potassium < 3.5 Or > 5.5 Meq/L)
* Patient With Symptomatic Heart Failure (Classes 3 And 4)
* Patient With A Prior Myocardial Infarction Or Stroke Within The Last 6 Months
* Patient Who Has Undergone Percutaneous Coronary Angioplasty Or Coronary Artery Bypass Within The Last 3 Months
* Pregnant Woman Or A Woman Of Childbearing Potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1738 (Actual)
Dates: Start 2005-09-01 (Actual); Primary Completion 2008-01-01 (Actual); Study Completion 2008-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Racine N, Hamet P, Sampalis JS, Longo N, Bastien N. A 52-week prospective, cohort study of the effects of losartan with or without hydrochlorothiazide (HCTZ) in hypertensive patients with metabolic syndrome. J Hum Hypertens. 2010 Nov;24(11):739-48. doi: 10.1038/jhh.2010.3. Epub 2010 Feb 11. PMID 20147971

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In: 12-Sep-2005 Last Patient In: 29-Dec-2006 Last Patient Last Visit: 31-Jan-08 Total number of Sites (General Practitioners and Family Physicians in Canada): 209
Pre-assignment Details: 24 patients not included in the Intention to Treat (ITT) analysis because they did not receive study medication and had no follow up visits. Total ITT population = 1714.
Groups:
- Losartan +/- Hydrochlorothiazide: Patients could be titrated up from Cozaar 50 mg to Cozaar 100mg to losartan 100 mg + Hydrochlorothiazide 12.5 mg and losartan 100mg/ Hydrochlorothiazide 25 mg, in sequence at any subsequent visits only if needed to obtain Blood Pressure under 140/90 mm Hg.
Period: Overall Study
Arm/Group | Losartan +/- Hydrochlorothiazide
Started | 1738
Week 4 | 1714
Week 8 | 1680
Week 12 | 1650
Week 32 | 1583
Week 52 | 1511
Completed | 1511
Not Completed | 227
Not completed — Adverse Event | 47
Not completed — Lost to Follow-up | 144
Not completed — Protocol Violation | 9
Not completed — Withdrawal by Subject | 20
Not completed — Non Compliance | 7

BASELINE CHARACTERISTICS:
Arm/Group | Losartan +/- Hydrochlorothiazide
Number analyzed (Participants) | 1714
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.93 (11.29)
Age, Customized [Number; unit: participants]
  <=45.00 | 326
  45.01 - 52.00 | 359
  52.01 - 58.00 | 356
  58.01 - 65.00 | 346
  >=65.00 | 326
  Missing | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 734
  Male | 980
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 1451
  Black | 32
  Asian | 200
  Native American | 11
  Other | 19
  Missing | 1
Body Mass Index [Mean (Standard Deviation); unit: Kg/m2] | 33.23 (5.59)
C-Reactive Protein [Mean (Standard Deviation); unit: mg/L] | 5.4 (8.8)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 90.54 (8.16)
Fasting Blood Glucose [Mean (Standard Deviation); unit: mmol/L] | 5.7 (0.7)
Heart Rate [Mean (Standard Deviation); unit: Beats per Minute (BPM)] | 75 (8.0)
Hemoglobin A1c [Mean (Standard Deviation); unit: Percent] | 5.71 (0.59)
High Density Lipoprotein-C [Mean (Standard Deviation); unit: mol/L] | 1.23 (0.33)
Low Density Lipoprotein-C [Mean (Standard Deviation); unit: mmol/L] | 3.17 (0.93)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 148.22 (10.72)
Total Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 5.36 (1.05)
Triglycerides [Mean (Standard Deviation); unit: mmol/L] | 2.16 (1.16)
Uric Acid [Mean (Standard Deviation); unit: mmol/L] | 365.8 (85.4)
Weight [Mean (Standard Deviation); unit: Kilograms (Kg)] | 92.5 (18.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1c Between 52 Weeks and Baseline
Description: Absolute Change in Hemoglobin A1c between 52 week measurement and baseline value.
Time Frame: 52 Weeks - Baseline
Population: Per Protocol
Measure: Median (Standard Deviation); unit: Percent
Groups:
- Losartan +/- Hydrochlorothiazide: Patients that completed 52 weeks of treatment and were >= 80% compliant with the study medication.
Arm/Group | Losartan +/- Hydrochlorothiazide
Number analyzed (Participants) | 1511
Percent | 0.04 (0.62)
Statistical Analysis 1: Comparison: Losartan +/- Hydrochlorothiazide; Single Cohort Study. Statistical Analysis is based on change from baseline. Null hypothesis value is + 0.5%; Test type: Superiority or Other; p = 0.999, t-test, 1 sided; Mean Difference (Final Values) = 0.02, 95% CI [-0.02 to 0.06], Standard Deviation 0.74

2. Primary Outcome: Change in Fasting Blood Glucose Between Baseline and 52 Weeks Assessments
Description: Absolute Change in Fasting Blood Glucose Measurements between Baseline and 52 week assessments.
Time Frame: 52 Weeks - Baseline
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Losartan +/- Hydrochlorothiazide
Number analyzed (Participants) | 1511
mmol/L | 0.02 (0.74)
Statistical Analysis 1: Comparison: Losartan +/- Hydrochlorothiazide; Single Cohort Study. Statistical Analysis is based on change from baseline. Null hypothesis value is + 0.5mmol/L; Test type: Superiority or Other; p = 0.999, t-test, 1 sided; Mean Difference (Final Values) = 0.04, 95% CI [0.01 to 0.07], Standard Deviation 0.62

3. Secondary Outcome: Target Blood Pressure
Description: Target Blood Pressure defined as Systolic Blood Pressure/Diastolic Blood Pressure ≤ 140/90 mm Hg at 52 weeks
Time Frame: 52 Weeks
Population: ITT and Per Protocol
Measure: Number; unit: Participants
Groups:
- Overall Total: All patients enrolled (signed the informed consent).
- Overall Intend to Treat: All patients enrolled and receiving at least one dose of study drug and having at least one follow up visit.
- Overall Per Protocol: All patients completing the 52 week study follow up.
Arm/Group | Overall Total | Overall Intend to Treat | Overall Per Protocol
Number analyzed (Participants) | 1738 | 1714 | 1511
Participants
  Achieved Target Blood Pressure | 1200 | 1200 | 1200
  Did NOT achieve target Blood Pressure | 538 | 514 | 311

4. Secondary Outcome: Change in Systolic Blood Pressure Between Baseline and 52 Week Assessments
Description: Absolute change in Systolic Blood Pressure between baseline and 52 week assessments.
Time Frame: 52 Weeks - Baseline
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Losartan +/- Hydrochlorothiazide
Number analyzed (Participants) | 1511
mm Hg | -16.95 (13.34)
Statistical Analysis 1: Comparison: Losartan +/- Hydrochlorothiazide; Single Cohort Study. Statistical Analysis is based on change from baseline. Null hypothesis value is 0 mm Hg; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -16.95, 95% CI [-17.62 to -16.27], Standard Deviation 13.34

5. Secondary Outcome: Change in Diastolic Blood Pressure Between Baseline and 52 Week Assessments
Description: Absolute change in Diastolic Blood Pressure between baseline and 52 week assessments.
Time Frame: 52 Weeks - Baseline
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Losartan +/- Hydrochlorothiazide
Number analyzed (Participants) | 1511
mm Hg | -9.84 (8.93)
Statistical Analysis 1: Comparison: Losartan +/- Hydrochlorothiazide; Single Cohort Study. Statistical Analysis is based on change from baseline. Null hypothesis value is 0 mm Hg; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -9.84, 95% CI [-10.29 to -9.39], Standard Deviation 8.39

6. Other Pre Specified Outcome: Change in Waist Circumference Between Baseline and 52 Week Assessments
Description: Absolute change in Waist Circumference between baseline and 52 week assessments
Time Frame: 52 Weeks - Baseline
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Losartan +/- Hydrochlorothiazide
Number analyzed (Participants) | 1511
cm | -1.28 (5.44)
Statistical Analysis 1: Comparison: Losartan +/- Hydrochlorothiazide; Single Cohort Study. Statistical Analysis is based on change from baseline. Null Hypothesis value is 0; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -1.3, Standard Deviation 5.4

7. Other Pre Specified Outcome: Change in Body Mass Index Between Baseline and 52 Week Assessments
Description: Absolute change in Body Mass Index Baseline and 52 week assessments
Time Frame: 52 Weeks - Baseline
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: Kg/m2
Arm/Group | Losartan +/- Hydrochlorothiazide
Number analyzed (Participants) | 1511
Kg/m2 | -7.3 (5.20)
Statistical Analysis 1: Comparison: Losartan +/- Hydrochlorothiazide; Single Cohort Study. Statistical Analysis is based on change from baseline. Null Hypothesis value is 0; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -7.3, Standard Deviation 5.20

8. Other Pre Specified Outcome: Percent Change in Low Density Lipoprotein-C Between Baseline and 52 Week Assessments
Description: Percent Change in LDL-C Between Baseline and 52 week assessments: 100% x [(LDL-C 52 Weeks - LDL-C Baseline) / (LDL-C Baseline)].
Time Frame: 52 Weeks - Baseline
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Losartan +/- Hydrochlorothiazide
Number analyzed (Participants) | 1511
Percent Change | -1.49 (32.10)
Statistical Analysis 1: Comparison: Losartan +/- Hydrochlorothiazide; Single Cohort Study. Statistical Analysis is based on change from baseline. Null Hypothesis value is 0; Test type: Superiority or Other; p = 0.084, t-test, 2 sided; Mean Difference (Net) = -1.5, Standard Deviation 32.1

9. Other Pre Specified Outcome: Percent Change in High Density Lipoprotein-C Between Baseline and 52 Week Assessments
Description: Percent Change in HDL-C Between Baseline and 52 week assessments: 100% x [(HDL-C 52 Weeks - HDL-C 52 Baseline) / (HDL-C Baseline)].
Time Frame: 52 Weeks - Baseline
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Losartan +/- Hydrochlorothiazide
Number analyzed (Participants) | 1511
Percent Change | 0.21 (17.96)
Statistical Analysis 1: Comparison: Losartan +/- Hydrochlorothiazide; Single Cohort Study. Statistical Analysis is based on change from baseline. Null Hypothesis value is 0; Test type: Superiority or Other; p = 0.654, t-test, 2 sided; Mean Difference (Final Values) = 0.2, Standard Deviation 18.0

10. Other Pre Specified Outcome: Percent Change in Triglycerides Between Baseline and 52 Week Assessments
Description: Percent Change in Triglycerides Between Baseline and 52 week assessments: 100% x [(Triglycerides 52 Weeks - Triglycerides Baseline) / (Triglycerides Baseline)].
Time Frame: 52 Weeks - Baseline
Population: Per Protocol
Measure: Median (Standard Deviation); unit: Percent Change
Arm/Group | Losartan +/- Hydrochlorothiazide
Number analyzed (Participants) | 1511
Percent Change | 1.09 (43.54)
Statistical Analysis 1: Comparison: Losartan +/- Hydrochlorothiazide; Single Cohort Study. Statistical Analysis is based on change from baseline. Null Hypothesis value is 0; Test type: Superiority or Other; p = 0.336, t-test, 2 sided; Mean Difference (Final Values) = -1.1, Standard Deviation 43.5

11. Other Pre Specified Outcome: Percent Change in Total Cholesterol Between Baseline and 52 Week Assessments
Description: Percent Change in Total Cholesterol Between Baseline and 52 week assessments: 100% x [(Total Cholesterol 52 weeks - Total Cholesterol Baseline) / (Total Cholesterol Baseline)].
Time Frame: 52 Weeks - Baseline
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Losartan +/- Hydrochlorothiazide
Number analyzed (Participants) | 1511
Percent Change | -2.98 (16.97)
Statistical Analysis 1: Comparison: Losartan +/- Hydrochlorothiazide; Single Cohort Study. Statistical Analysis is based on change from baseline. Null Hypothesis value is 0; Test type: Superiority or Other; p = 0.001, t-test, 2 sided; Mean Difference (Final Values) = -3.0, Standard Deviation 17.0

12. Other Pre Specified Outcome: Absolute Change in Uric Acid Between Baseline and 52 Week Assessments
Description: Absolute Change in Uric Acid Between Baseline and 52 week assessments: Uric Acid 52 weeks - Uric Acid Baseline.
Time Frame: 52 Weeks - Baseline
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Losartan +/- Hydrochlorothiazide
Number analyzed (Participants) | 1511
mmol/L | -19.17 (63.84)
Statistical Analysis 1: Comparison: Losartan +/- Hydrochlorothiazide; Single Cohort Study. Statistical Analysis is based on change from baseline. Null Hypothesis value is 0; Test type: Superiority or Other; p = 0.001, t-test, 2 sided; Mean Difference (Final Values) = -19.2, Standard Deviation 63.8

13. Other Pre Specified Outcome: Absolute Change in C Reactive Protein Between Baseline and 52 Week Assessments
Description: Absolute Change in C Reactive Protein Between Baseline and 52 week assessments: C Reactive Protein 52 weeks - C Reactive Protein Baseline.
Time Frame: 52 Weeks - Baseline
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Losartan +/- Hydrochlorothiazide
Number analyzed (Participants) | 1511
mg/L | -0.36 (8.66)
Statistical Analysis 1: Comparison: Losartan +/- Hydrochlorothiazide; Single Cohort Study. Statistical Analysis is based on change from baseline. Null Hypothesis value is 0; Test type: Superiority or Other; p = 0.613, t-test, 2 sided; Mean Difference (Final Values) = -0.4, Standard Deviation 8.7

ADVERSE EVENTS:
Arm/Group | Overall ITT
Serious Adverse Events (participants affected / at risk) | 35/1714
Other Adverse Events (participants affected / at risk) | 198/1714
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall ITT (N=1714)
Acute coronary syndrome (Cardiac disorders) | 1
Acute depression (Psychiatric disorders) | 1
Acute renal insufficiency (Renal and urinary disorders) | 1
Anaphylactic shock (Immune system disorders) | 1
Anaphylaxis (Immune system disorders) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Atherosclerotic cardiovascular disease (Vascular disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Bronchitis asthmatic (Respiratory, thoracic and mediastinal disorders) | 1
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Cardiac catheterization (Surgical and medical procedures) | 1
Cardiomyopathy (Cardiac disorders) | 1
Cerebral vascular accident (Nervous system disorders) | 3
Chest Pain (General disorders) | 1
Death (General disorders) | 2
Gastric Ulcer (Gastrointestinal disorders) | 1
Hip Replacement (Surgical and medical procedures) | 2
Ileostomy (Surgical and medical procedures) | 1
Infarction (Cardiac disorders) | 1
Lymphoma grade IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Multiple sclerosis aggravated (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Numbness of Upper Arm (Nervous system disorders) | 1
Pneumonia (Infections and infestations) | 1
Rotator Cuff Repair (Surgical and medical procedures) | 1
Single Vessel Disease (Cardiac disorders) | 1
Subarachnoid Hemorrhage (Nervous system disorders) | 1
Superficial Femoral Arterial Stenosis (Vascular disorders) | 1
Ulcer Bleeding Gastric (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Overall ITT (N=1714)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 54
Dizziness (Nervous system disorders) | 35
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 29
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 23
Headache (Nervous system disorders) | 21
Sinusitis (Infections and infestations) | 19
Blood Glucose Increased (per investigator's clinical judgment) (Investigations) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.